CLINICAL TRIAL: NCT01540942
Title: A Randomized, Controlled, Open-label Study to Investigate the Impact of Disease Activity and Nutrition Treat on Postoperative Recurrence and Complications After Bowel Resection for Crohn's Disease
Brief Title: Impact of Disease Activity and Nutrition Treat on Postoperative Recurrence and Complications After Bowel Resection for Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Zhu Weiming, vice director of General surgery institute, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDS-1
Record Dates: First submitted 2012-02-23; First posted 2012-02-29 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Nutrition; Bowel resection; Postoperative recurrence; complication; Active disease
MeSH Terms: conditions — Crohn Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Nutrition treat (Active Comparator): perioperative nutrition support until the patients get the normal nutrition or disease remission
  Interventions: Dietary Supplement: nutrition treat
- bowel resection (Active Comparator): bowel resection until the patients get the normal nutrition or disease remission after bowel resection
  Interventions: Other: surgery

INTERVENTIONS:
Dietary Supplement: nutrition treat — intestinal nutrition treat :female：REE（Kcal/d）=655+9.6W+1.7H-4.7A; male：REE（Kcal/d）=66+13.7W+5.0H-6.8A;[W=weight（Kg）；H=height（cm）；A=age（year）]
  Arms: Nutrition treat
Other: surgery — bowel resection
  Arms: bowel resection

SUMMARY:
The study was aimed to determine whether perioperative nutrition treat and(or)the perioperative disease activity were associated with postoperative recurrence and complications after bowel resection for Crohn's disease.

DETAILED DESCRIPTION:
The investigators want to assess the impact of possible risk factors on intestinal resection and postoperative recurrence in Crohn's disease (CD) and to evaluate the disease course.

In our clinical treatments, the investigators found that perioperative CDAI and nutrition treatment may have same impact on postoperative recurrence and complication in Crohn's disease. The investigators design this study to test it.

The study prepare to collect the clinical data of patients who need bowel resection for CD to analyzed. The investigators divide those patients into two groups (N,I group). They accept intestinal nutrition with the respective aim that get the inflammatory index (erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), Crohns Disease Activity Index (CDAI)) norm or nutritional index norm before they accept surgery. Postoperative recurrence and complications in patients will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

Patients had a CRP level of more than 8mg/L Patients had a preoperative weight loss >5% over the past 6 months and had a serum albumin of less than 35g/L at the enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 4 weeks

SECONDARY OUTCOMES:
postoperative recurrence | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Weiming Zhu, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Olaison G, Smedh K, Sjodahl R. Natural course of Crohn's disease after ileocolic resection: endoscopically visualised ileal ulcers preceding symptoms. Gut. 1992 Mar;33(3):331-5. doi: 10.1136/gut.33.3.331. PMID 1568651
- [Background] Reese GE, Nanidis T, Borysiewicz C, Yamamoto T, Orchard T, Tekkis PP. The effect of smoking after surgery for Crohn's disease: a meta-analysis of observational studies. Int J Colorectal Dis. 2008 Dec;23(12):1213-21. doi: 10.1007/s00384-008-0542-9. Epub 2008 Sep 2. PMID 18762954
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Rutgeerts P, Geboes K, Vantrappen G, Kerremans R, Coenegrachts JL, Coremans G. Natural history of recurrent Crohn's disease at the ileocolonic anastomosis after curative surgery. Gut. 1984 Jun;25(6):665-72. doi: 10.1136/gut.25.6.665. PMID 6735250
- [Background] McLeod RS, Wolff BG, Ross S, Parkes R, McKenzie M; Investigators of the CAST Trial. Recurrence of Crohn's disease after ileocolic resection is not affected by anastomotic type: results of a multicenter, randomized, controlled trial. Dis Colon Rectum. 2009 May;52(5):919-27. doi: 10.1007/DCR.0b013e3181a4fa58. PMID 19502857
- [Background] Yamamoto T. Factors affecting recurrence after surgery for Crohn's disease. World J Gastroenterol. 2005 Jul 14;11(26):3971-9. doi: 10.3748/wjg.v11.i26.3971. PMID 15996018
- [Background] Cosnes J, Beaugerie L, Carbonnel F, Gendre JP. Smoking cessation and the course of Crohn's disease: an intervention study. Gastroenterology. 2001 Apr;120(5):1093-9. doi: 10.1053/gast.2001.23231. PMID 11266373
- [Background] Johnson GJ, Cosnes J, Mansfield JC. Review article: smoking cessation as primary therapy to modify the course of Crohn's disease. Aliment Pharmacol Ther. 2005 Apr 15;21(8):921-31. doi: 10.1111/j.1365-2036.2005.02424.x. PMID 15813828
- [Derived] Zhu W, Guo Z, Zuo L, Gong J, Li Y, Gu L, Cao L, Li N, Li J. CONSORT: Different End-Points of Preoperative Nutrition and Outcome of Bowel Resection of Crohn Disease: A Randomized Clinical Trial. Medicine (Baltimore). 2015 Jul;94(29):e1175. doi: 10.1097/MD.0000000000001175. PMID 26200619